CLINICAL TRIAL: NCT01231386
Title: MIRNA Profiling of Breast Cancer in Patients Undergoing Neoadjuvant or Adjuvant Treatment for Locally Advanced & Inflammatory Breast Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09147
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Female Breast Cancer; miRNA expression; Neoadjuvant/Adjuvant Treatment; Locally and Inflammatory Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue and Blood Procurement. Breast cancer tissues from core biopsies (as available, preferably fresh frozen or RNA-later preserved, but in case of lack of availability, formalin-fixed paraffin-embedded [FFPE] core or tissue samples) which have been collected or will be collected under IRB#05091 or 05015.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
MicroRNAs (MiRNAs) regulate the translation of RNAs and are implicated in cell proliferation and renewal both under physiologically normal as well as in malignant conditions. Dysregulation of specific miRNAs may be associated with either gaining oncogenic or loosing tumor suppressing functions. MiRNA dysregulation has been implicated in breast cancer tumorigenic (stem cell) and non-tumorigenic development. Therefore, miRNA profiling of treatment naïve and treatment-exposed breast tumors and sequential samples of blood/serum will allow for identification of miRNA markers of prognosis and as indicators and potential targets for personalized therapies. In this proposal, specimens from patients treated in the clinical breast cancer program on already existing protocols (IRB 05091 and 05015) will be characterized by Dr. Rossi's laboratory and collaborators, and the information gained will be applied to develop specific therapies.

DETAILED DESCRIPTION:
Current neoadjuvant or adjuvant treatment strategies do not allow for rationale incorporation of such agents. One needs tools to predict both de novo and acquired resistance to therapeutic agents. This is a difficult task, due to the compound nature of escape routes: tumor exposure is usually to a combination of therapeutic agents and the mechanisms of resistance are broad: intrinsic resistance due to existing mutations, or regulatory - miRNA, other epigenetic - alterations, polymorphisms, tumor cell adaptation via new mutations and activation of alternative pathways, lack of optimal pharmacokinetics/genomics, activation of efflux mechanisms, accelerated repair mechanisms are involved.

Similarly, not all patients who are candidates for primary surgical intervention to be followed by post-operative adjuvant therapy benefit from such systemic treatments. The mechanisms of resistance be it de novo in surviving stem cell/tumorigenic components, or acquired by cells left behind "dormant" after the surgical intervention, are not well delineated.

Breast tumors subjected to neoadjuvant chemotherapy allow for baseline and treatment-effected sampling. Characterization of core biopsy specimens of primary tumors procured prior to exposure to neoadjuvant therapy from different varieties of breast cancer subtypes, and of subsequent mid-treatment and intraoperative (procured during definitive surgery following completion of neoadjuvant therapy) samples should help to assess the predictive value of the pre-treatment and post-treatment miRNA expression profile for complete and near complete response, as a surrogate marker for survival. Similarly, patterns of de novo and acquired resistance may emerge when assessment of pre- and post treatment miRNA expression profiles are analyzed in a supervised manner of classification using pathological response as classifier. Samples obtained from patients with primary surgical removal of their tumors before any systemic treatment exposure on the other hand, will allow for determining markers of prognosis, and predictors for response to therapeutic targeting agents.

Time Perspective: Retrospective/Prospective

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Breast Cancer
* > 18 years,
* regardless of histology, treatment phase, or stage

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female, Breast Cancer, > 18 years, regardless of histology, treatment phase, or stage. However, only patients with Stage II-III disease from IRB #05015 will be accrued, in order to assure that sufficient tumor tissue will be available.
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2009-11; Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Performance of miRNA profiling from tumor samples from primary breast tumors | 3 years after completion of sample collection
Assessment of miRNA profiles from blood/serum samples from patients at baseline, and if feasible, at different time points | 3 years after completion of sample collection
Analysis of miRNA findings and correlate miRNA patterns of expression in tumor, lymph nodes -if available- and in serum | 3 years after competion of sample collection
Correlation of classic tumor markers such as estrogen and progesterone receptor (ER,PR), and HER2 expression with tumor stage and grade | 3 years after completion of sample collection
Determination of specific miRNA functions | 3 years after completion of sample collection
Determination of ability to knock down functionally relevant overexpressed miRNAs by miR-sponge/antagomirs | 3 years after completion of sample collection
Design of prospective pilot phase I-II trials to interfere with dysfunctional/dysregulated miRNA expression | 3 years after completion of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States